CLINICAL TRIAL: NCT01544426
Title: Does Office Hysteroscopy and Endometrial Snip Improve IUI Outcome? : a Randomized Controlled Trial
Brief Title: Office Hysteroscopy and Endometrial Snip Improve Intrauterine Insemination Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42012
Record Dates: First submitted 2012-02-26; First posted 2012-03-06 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
Keywords: Office hysteroscopy,; intrauterine insemination; endometrial scrap
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Office hysteroscopy and endometrial snip (Experimental): Office hysteroscopy and endometrial snip
  Interventions: Procedure: Office hysteroscopy and endometrial snip
- Office hyteroscopy (Active Comparator): Office hysteroscopy
  Interventions: Procedure: Office hysteroscopy

INTERVENTIONS:
Procedure: Office hysteroscopy and endometrial snip — Office hysteroscopy with endometrial snip
  Other Names: Office hysteroscopy combined with endometrial snip
  Arms: Office hysteroscopy and endometrial snip
Procedure: Office hysteroscopy — Office hysteroscopy
  Other Names: Outpatient hysteroscopy
  Arms: Office hyteroscopy

SUMMARY:
Endometrial injury had been studied before prior to intracytoplasmic sperm injection (ICSI) cycles , in cases of repeated implantation failure. It is found that it will improve the implantation rate.

DETAILED DESCRIPTION:
The investigators can combine office hysteroscopy to diagnose hidden endometrial pathology, with hysteroscopically guided endometrial snip from the fundus of the uterus, trying to improve the pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* 18- 38 years old
* at least one patent tube
* unexplained infertility, anovulation, mild to moderate male factor infertility
* previous failed IUI

Exclusion Criteria:

* indicated for ICSI

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 332 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 10 month
  Positive pregnancy test with fetal heart activity

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 12 month
  Pregnancy Continued after 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khayat, M.D., Principal Investigator — Cairo University
Locations (1):
- Kasr Al-AINY hospital, Cairo, Egypt

REFERENCES:
- [Derived] El-Khayat W, Elsadek M, Saber W. RETRACTED: Comparing the effect of office hysteroscopy with endometrial scratch versus office hysteroscopy on intrauterine insemination outcome: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:96-100. doi: 10.1016/j.ejogrb.2015.08.025. Epub 2015 Aug 28. PMID 26344351 (Retraction: PMID 35870425 Eur J Obstet Gynecol Reprod Biol. 2022 Sep;276:118)